CLINICAL TRIAL: NCT04058496
Title: The Importance of Wnt-signaling in the Pathobiology of Systemic Inflammation and Organ Dysfunction After Cardiac Surgery
Brief Title: The Importance of Wnt-signaling After Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Alain Rudiger (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor-Investigator, Alain Rudiger, Prof. Dr. med., University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: Wnt-study
Record Dates: First submitted 2019-06-21; First posted 2019-08-15 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Inflammation; Thoracic Surgery
Keywords: Cardia surgery; Cardio-pulmonary bypass; Inflammation; WNT; Cytokines
MeSH Terms: conditions — Inflammation | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: Coronary artery bypass surgery off-pump (n=24)
  Interventions: Other: Blood sampling
- 2: Coronary artery bypass surgery on-pump (n=16)
  Interventions: Other: Blood sampling
- 3: Coronary artery bypass surgery plus valve surgery (n=20)
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Five Timepoints: baseline (pre-operative), ICU admission, 4 hours after ICU admission, 8 hours after ICU admission, 48 hours after ICU admission

SUMMARY:
Cardiac surgery saves lives when patients suffer from cardiac disease. Local inflammation is important for tissue repair and wound healing after such an operation. Inflammation starts already when the patient is treated in the intensive care unit. When inflammatory proteins (cytokines) are released into the circulation, they cause also a systemic inflammation, which alerts the immune system of the body and activates defence mechanisms (=adaptive response). In some patients, systemic inflammation is out of control thereby causing organ dysfunctions, shock, and in the most severe cases even death (=maladaptive response). The aim of this study is to investigate the early phase of inflammation after the operation. Repeated blood samples will be taken of patients undergoing cardiac surgery to describe the patterns and dynamics of inflammation proteins. A better understanding of these mechanisms will potentially lead to improved treatment of patients after cardiac surgery.

DETAILED DESCRIPTION:
The aim of this project is to understand early inflammation mechanisms after cardiac surgery. Therefore, repeated blood samples of patients undergoing cardiac surgery will be taken. Patients are selected after "open" cardiac surgery (via sternotomy), when when they require postoperative care in the cardiovascular intensive care unit. The blood samples will be analysed in collaboration with the Inflammation Research Unit of the Department of Internal Medicine at the University Hospital Zurich.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery via sternotomy
* Coronary-bypass bypass surgery with or without valve surgery
* Postoperative hospitalisation in the cardio-surgical ICU
* Available informed consent

Exclusion Criteria:

* Preoperative infections (e.g. endocarditis)
* Preoperative use of steroids or other immunosuppression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after open cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of Wnt5a (ng/ml) | Up to 48 hours after ICU admission
  Measured by a commercially available ELISA
Plasma concentration of sFRP1 (ng/ml) | Up to 48 hours after ICU admission
  Measured by a commercially available ELISA
Plasma concentration of sFRP5 (ng/ml) | Up to 48 hours after ICU admission
  Measured by a commercially available ELISA
Plasma concentration of WIF-1 (pg/ml) | Up to 48 hours after ICU admission
  Measured by a commercially available ELISA

SECONDARY OUTCOMES:
Daily fluid balance (ml) | Up to 48 hours after ICU admission
  Routine parameter taken from charts
Occurrence of complications (yes/no): composite endpoint of hemodynamic instability (defined as norepinephrine concentration = or > 0.1mcg/kg/min), delirium (defined as ICDSC score = or > 4), infections | Up to 7 days after ICU admission
  Routine parameter taken from charts
Length of ICU stay (days) | Up to 4 weeks
  Routine parameter taken from charts

CONTACTS AND LOCATIONS:
Overall Officials: Alain Rudiger, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital, Zurich, Switzerland

REFERENCES:
- [Background] Hauffe T, Kruger B, Bettex D, Rudiger A. Shock Management for Cardio-surgical ICU Patients - The Golden Hours. Card Fail Rev. 2015 Oct;1(2):75-82. doi: 10.15420/cfr.2015.1.2.75. PMID 28785436
- [Background] Hauffe T, Kruger B, Bettex D, Rudiger A. Shock Management for Cardio-surgical Intensive Care Unit Patient: The Silver Days. Card Fail Rev. 2016 May;2(1):56-62. doi: 10.15420/cfr.2015:27:2. PMID 28785454
- [Derived] Kruger BD, Hofer GE, Rudiger A, Spahn GH, Braun J, Bettex D, Schoedon G, Spahn DR. Wingless-related integration site (WNT) signaling is activated during the inflammatory response upon cardiac surgery: A translational study. Front Cardiovasc Med. 2022 Nov 11;9:997350. doi: 10.3389/fcvm.2022.997350. eCollection 2022. PMID 36440011